CLINICAL TRIAL: NCT07029321
Title: Effect of Modified Poco-Poco Exercise to Tongue Strength, Cognitive Function and Quality of Life in Elderly
Brief Title: Effect of Modified Poco-Poco Exercise to Cognitive Function and Quality of Life in Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Irma Ruslina Defi, Principal Investigator, Universitas Padjadjaran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKFR.1103.06.25
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Geriatrics Rehabilitation

STUDY DESIGN:
Intervention Model Description: Modified poco-poco exercises
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified poco-poco exercises (Experimental): Participants performed modified poco-poco exercise program for 12 weeks and were assessed tongue strength, cognitive function, and quality of life
  Interventions: Procedure: Modified poco-poco exercises

INTERVENTIONS:
Procedure: Modified poco-poco exercises — Participants performed modified poco-poco exercises for 12 weeks

SUMMARY:
Subjects with sarcopenia will get a modified poco-poco exercise program was assessed for tongue strength, cognitive function, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years old or above
* Have sarcopenia (based on AWGSOP 2019 criteria)
* MoCA INA score 18 - 25
* Tongue strength < 35 kPa

Exclusion Criteria:

* Hearing impairment/loss hindering participants to receive verbal instructions
* Vision impairment/loss hindering participants to receive instructions
* Musculoskeletal impairment hindering participants to do exercise
* Participants have been involved in other exercise program
* Severe joint diseases
* Severe cardiovascular disease diagnosed by Cardiologist Previous dysphagia oropharyngeal caused by anatomical and or neuromuscular diseases
* Front dental loss

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Tongue Strength | 12 weeks
  Tongue strength will be assessed by Maximum Isometric Pressure (MIP) - score in kilopascal
Cognitive Function | 12 weeks
  Cognitive Function will be assessed by Montreal Cognitive Assessment Indonesian Version (MoCA-Ina) - score in numerical 0-30
Quality of Life using a questionnaire | 12 weeks
  Quality of Life will be assessed by Sarcopenia and Quality of Life Questionnaire (SARQOL) - score in numerical 0-100